CLINICAL TRIAL: NCT03218813
Title: A Pharmacist-Led Hospital-Based Intervention to Support Medication Adherence Following Acute Coronary Syndrome: An Intervention Cohort Study
Brief Title: A Pharmacist-Led Hospital-Based Intervention to Support Medication Adherence Following Acute Coronary Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: v1 30-06-17
Record Dates: First submitted 2017-07-12; First posted 2017-07-17 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2018-08

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Intervention Model Description: This study will adopt a non-randomised prospective intervention cohort design (i.e. controlled before-and-after (CBA) study). Two cohorts of patients will be recruited from a single NHS site over two recruitment periods. Pharmacists will be trained between these recruitment periods to deliver an intervention, thus creating two comparable groups (control/'before' group vs. intervention/'after' group).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control cohort ('before' group) (No Intervention): Control cohort ('before' group): eligible patients will receive treatment as usual (TAU) and will complete all outcome measures.
- Intervention cohort ('after' group) (Experimental): Eligible patients will receive the pharmacist-led intervention and will complete all outcome measures.
  Interventions: Behavioral: Intervention cohort ('after' group)

INTERVENTIONS:
Behavioral: Intervention cohort ('after' group) — The intervention will take place during hospitalisation. Patients will complete the BMQ-S and their responses will form the basis of what will be discussed in Session 1. Pharmacists will elicit patients' thoughts and opinions about their medicines and highlight the need to take them. Any erroneous treatment beliefs will be discussed and any concerns will be addressed.
  After Session 1, patients will be given a planning sheet and will be asked to think about their usual daily routine and how taking medicines may fit into it. Session 2 will focus on developing specific action plans for taking medication at home. Patients will be asked to formulate an if-then plan ('If it is time X in place Y and I am doing Z, then I will take my pill dose').
  Arms: Intervention cohort ('after' group)

SUMMARY:
Background Medication adherence following acute coronary syndrome (ACS) is often sub-optimal and is associated with poor clinical outcomes. Patients' beliefs about medications have been shown to predict poor adherence and may be targetable for intervention. Findings novel ways to improve adherence is an important area of research with widespread clinical implications. Pharmacists may currently be underutilised in promoting and monitoring medication-taking behaviour. There have been few effective interventions led by pharmacists to support medication adherence in patients with ACS.

Objectives This study follows on from a feasibility and acceptability study recently conducted (NCT02967588). The primary objective is to pilot a pharmacist-led hospital-based intervention to support medication adherence following an ACS.

Methods This study will adopt a non-randomised intervention cohort design (i.e. controlled before-and-after (CBA) study). Patients admitted to hospital with an ACS will be recruited for this study. Patients must be prescribed medicines for secondary prevention. The study will be delivered by hospital pharmacists over two sessions and will target both intentional (Session 1) and unintentional (Session 2) adherence barriers. Session 1 will involve eliciting and challenging patients' erroneous beliefs about medications. Session 2 will involve formulating specific action plans to encourage medication-taking habit formation.

Outcome Outcome data will be collected at two time points - 6 week and 12 week follow up. The primary outcome of this proposed study will be treatment beliefs, measured using the Beliefs about Medicines Questionnaire-Specific (BMQ-S) (Horne, Weinman & Hankin, 1999). Our secondary outcome will be self-reported medication adherence measured using the Medication Adherence Report Scale (MARS-5) (Horne & Weinman, 2002). Depression, medicines-related self-efficacy and satisfaction with medicines information provision will also be measured.

Study timeline Control cohort ('before' group): eligible patients will receive treatment as usual (TAU) and will complete all outcome measures (i.e. treatment beliefs, medication adherence). Pharmacists will then be trained to deliver the intervention. Intervention cohort ('after' group): eligible patients will receive the pharmacist-led intervention and will complete all outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and over
* Clinical diagnosis of ACS*
* ACS primary reason for hospitalisation
* Patients to be prescribed medications for secondary prevention (i.e. antiplatelet drugs, statins, ACEi, ARBs, β-blockers)
* Sufficient spoken English to participate in the study

Exclusion Criteria:

* Under 18 years of age
* Developed ACS* as a secondary condition (i.e. perioperative MI)
* Not prescribed medications for secondary prevention (i.e. antiplatelet drugs, statins, ACEi, ARBs, β-blockers)
* Non-English speaking
* Medical notes indicate cognitive impairment

  *ACS is defined as patients diagnosed with a myocardial infarction or unstable angina (European Society of Cardiology Clinical Practice Guidelines (Roffi et al., 2015; Steg et al., 2012)).
* Non-ST-segment elevated myocardial infarction (NSTEMI) - Myocardial ischaemia with elevated cardiac biomarkers (i.e. troponin) in the absence of ST-segment elevation identified via electrocardiogram (ECG).
* ST-segment elevated myocardial infarction (STEMI) - Myocardial ischaemia with elevated cardiac biomarkers (i.e. troponin) and ST-segment elevation identified via electrocardiogram (ECG).
* Unstable angina - Myocardial ischaemia at rest or minimal exertion in the absence of cardiomyocyte necrosis and significantly elevated cardiac biomarkers (i.e. troponin).

All diagnoses will be made by the patients' clinical team. The research team will play no part in this process.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2017-12-12 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Treatment beliefs | 12 week follow up
  Beliefs about Medication Questionnaire-Specific (BMQ-S)

SECONDARY OUTCOMES:
Treatment beliefs | 6 week follow up
  Beliefs about Medication Questionnaire-Specific (BMQ-S)
Medication adherence | 12 week follow up
  Medication Adherence Report Scale-5 (MARS-5)
Medication adherence | 6 week follow up
  Medication Adherence Report Scale-5 (MARS-5)
Depression | 12 week follow up
  Patient Health Questionnaire-2 (PHQ-2)
Medicines-related self-efficacy | 12 week follow up
  Self-Efficacy for Appropriate Medication Use Scale (SEAMS)

CONTACTS AND LOCATIONS:
Locations (1):
- Guy's & St Thomas' NHS Foundation Trust, London, United Kingdom